CLINICAL TRIAL: NCT03115632
Title: Contributing Factors in the Pathobiology of Airway Remodeling in Obesity
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00077482
Record Dates: First submitted 2017-04-04; First posted 2017-04-14 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-06

CONDITIONS: Asthma; Obesity; Obesity, Morbid; Bariatric Surgery Candidate
MeSH Terms: conditions — Asthma; Obesity; Obesity, Morbid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood plasma, bronchoscopy with endobronchial biopsy and brushings, bronchoalveolar lavage, RNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Obese asthmatic & lean asthmatic: men and women with asthma and either obese or lean BMI
- Obese non-asthmatic & lean non-asthmatic: men and women without asthma and either obese or lean BMI
- Asthmatic undergoing bariatric surgery: Obese asthmatic men and women undergoing bariatric surgery
- Non-asthmatic undergoing bariatric surgery: Obese men and women undergoing bariatric surgery

SUMMARY:
There are two aims for this study. The purpose of this study is to determine the effects of body weight and hormones on airway fibrosis (scarring) and lung function in obese & lean asthma subjects compared to obese & lean non-asthma subjects (Aim 1). And in obese subjects with asthma undergoing bariatric surgery compared to obese non-asthma subjects undergoing bariatric surgery (Aim 2).

DETAILED DESCRIPTION:
Main Study

Specific Aim 1: Determine the effects of signaling on airway fibrosis and lung function in obese asthma and non-asthma patients. The investigators will:

•Perform assessments to determine if obese, early-onset asthma patients are more susceptible to airway fibrosis and remodeling than lean, early-onset asthma patients and obese and lean, non-asthma patients.◦

Specific Aim 2: Investigate the mechanism by which bariatric surgery slows the progression of airway fibrosis in obese human asthma. The investigators will:

•Perform assessments to determine if airway fibrosis in obese, early-onset asthma and obese non-asthma patients improves following bariatric surgery and weight loss◦

ELIGIBILITY:
Inclusion Criteria:

Obese asthmatic & lean asthmatic

1. Outpatient adults of either sex 18-60 years of age with an initial asthma diagnosis at < 12 years of age, as defined by the NHLBI National Asthma Education and Prevention Program (NAEPP) guidelines.
2. Lean subjects with body mass index (BMI) ≥ 20 kg/m2 and < 30 kg/m2 or obese subjects with BMI ≥ 30 and ≤ 55 kg/m2
3. Physician diagnosis of asthma
4. Forced expiratory volume at one second (FEV1) within acceptable limits (>45% predicted before and >55% predicted after, bronchodilator administration).
5. Negative pregnancy test in women of childbearing potential (confirmed during screening).
6. Relatively healthy subjects able to undergo bronchoscopy without complications.
7. Willing and able to give informed consent and adhere to visit/protocol schedules.
8. Read and write in English.

Obese non-asthmatic & Lean non-asthmatic

1. Outpatient adults of either sex 18-60 years of age.
2. Lean subjects with body mass index (BMI) ≥ 20 kg/m2 and < 30 kg/m2 or obese subjects with BMI ≥ 30 and ≤ 55 kg/m2
3. Negative pregnancy test in women of childbearing potential (confirmed during screening).
4. Normal lung function.
5. No clinical history of atopy.
6. No significant medical or psychological issues.
7. Healthy subjects able to undergo bronchoscopy without complications.
8. Willing and able to give informed consent and adhere to visit/protocol schedules.
9. Read and write in English.

Asthmatic undergoing bariatric surgery

1. Outpatient adults of either sex 18-60 years of age with an initial asthma diagnosis at < 12 years of age, as defined by the NHLBI NAEPP guidelines.
2. Physician diagnosis of asthma
3. FEV1 within acceptable limits (>45% predicted before and >55% predicted after, bronchodilator administration).
4. Morbidly obese subjects undergoing bariatric surgery and receiving care at the Duke Metabolic and Weight Loss Surgery Center.
5. Negative pregnancy test in women of childbearing potential (confirmed during screening).
6. Relatively healthy subjects able to undergo bronchoscopy without complications.
7. Willing and able to give informed consent and adhere to visit/protocol schedules.
8. Read and write in English.

Non-Asthmatic undergoing bariatric surgery

1. Outpatient adults of either sex 18-60 years of age.
2. Morbidly obese subjects undergoing bariatric surgery and receiving care at the Duke Metabolic and Weight Loss Surgery Center.
3. Negative pregnancy test in women of childbearing potential (confirmed during screening).
4. Normal lung function.
5. No clinical history of atopy.
6. No significant medical or psychological issues.
7. Healthy subjects able to undergo bronchoscopy without complications.
8. Willing and able to give informed consent and adhere to visit/protocol schedules.
9. Read and write in English.

Exclusion Criteria:

1. Children < 18 years of age.
2. Adults ≥ 18 years of age with an initial asthma diagnosis at ≥ 12 years of age, as defined by the NHLBI NAEPP guidelines.
3. Inpatient status.
4. FEV1 is less than 45% predicted before, or less than 55% predicted after, bronchodilator administration.
5. Upper or lower respiratory tract infection within one month of the study.
6. Use of inhaled or systemic corticosteroids within four weeks of study.
7. Use of long-acting beta-2, GLP-1 receptor agonists, or dipeptidyl peptidase-4 (DPP-4) inhibitors within two weeks of study.
8. Smoking history > 5 pack years or any cigarette use within the previous six months.
9. Significant non-asthma pulmonary disease (stable obstructive sleep apnea is not excluded).
10. Positive pregnancy test for women and/or nursing women.
11. An emergency department visit or inpatient admission for a primary respiratory diagnosis or treatment with antibiotics within 60 days of enrollment.
12. Poorly controlled concomitant conditions that pose additional procedure risk as determined by the investigator.
13. All patients on anticoagulants
14. Uncontrolled sleep apnea
15. Use of e-cigarettes or "vape" devices of any kind

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects will be recruited from the clinics of the Duke Asthma, Allergy and Airway Center, the Duke Metabolic and Weight Loss Surgery Center, the Duke Raleigh Weight Loss Surgery Center, and the Duke Diet and Fitness Center. Healthy controls without lung disease will be recruited from the surrounding area.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-06-27 (Actual)

PRIMARY OUTCOMES:
Airway fibrosis | Visit 2 (14 days)
  Obese asthmatics compared to lean asthmatics, obese non-asthmatics and lean non-asthmatics: A univariate linear model will be constructed to measure the effect of leptin or GLP-1 (glucagon-like peptide-1) on airway fibrosis, as measured by the ratio of Masson's trichrome-stained area to non-stained area in the sub-mucosal region of airway biopsy tissue.
Change in airway fibrosis | Visit 2 (14 days), Visit 4 (1 year + 14 days)
  Asthmatics undergoing bariatric surgery and non-asthmatics undergoing bariatric surgery: Each patient will serve as its own control in comparing pre- and post-operative airway fibrosis. A univariate linear model will be constructed to measure the effect of bariatric surgery on airway fibrosis, as measured by the ratio of Masson's trichrome-stained area to non-stained area in the sub-mucosal region of airway biopsy tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Loretta Que, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Duke Metabolic and Weight Loss Surgery Center, Durham, North Carolina
  - Duke Asthma Allergy and Airway Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No